CLINICAL TRIAL: NCT01505127
Title: A Phase 3, Randomized, Double-Blind, Double Dummy, Multicenter, Parallel Group Comparison Study to Evaluate Efficacy and Safety of a Triple Therapy With TAK-438, Amoxicillin and Clarithromycin by Comparison With a Triple Therapy With AG-1749 (Lansoprazole), Amoxicillin and Clarithromycin for the First Line Eradication of H.Pylori
Brief Title: Efficacy of TAK-438, Amoxicillin and Clarithromycin in the First Line Eradication of H. Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CCT-401; U1111-1126-5073 (Registry Identifier: WHO); JapicCTI-111722 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-12-30; First posted 2012-01-06 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: H. Pylori Infection
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-438 20 mg BID (Experimental): TAK-438 20 mg, tablets, orally, twice daily for 1 week
  Lansoprazole placebo-matching capsules, orally, twice daily for 1 week
  Amoxicillin 750 mg, capsules, orally, twice daily for 1 week
  Clarithromycin 200 or 400 mg, tablets, orally, twice daily for 1 week
  Interventions: Drug: TAK-438; Drug: Amoxicillin; Drug: Clarithromycin
- Lansoprazole 30 mg BID (Experimental): TAK-438 placebo-matching tablets, orally, twice daily for 1 week
  Lansoprazole 30 mg, capsules, orally, twice daily for 1 week
  Amoxicillin 750 mg, capsules, orally, twice daily for 1 week
  Clarithromycin 200 or 400 mg, tablets, orally, twice daily for 1 week
  Interventions: Drug: Lansoprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: TAK-438
  Arms: TAK-438 20 mg BID
Drug: Lansoprazole
  Other Names: AG-1749
  Arms: Lansoprazole 30 mg BID
Drug: Amoxicillin
Drug: Clarithromycin

SUMMARY:
The purpose of this study is to confirm the efficacy of triple therapy with TAK-438, Amoxicillin and Clarithromycin, twice daily (BID) by demonstrating its non-inferiority to triple therapy with Lansoprazole, Amoxicillin and Clarithromycin in H. pylori-positive patients with scarred gastric or duodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be H. pylori-positive patients at baseline (Visit 1)
2. Participants must be endoscopically confirmed to have scarred gastric ulcer or duodenal ulcer at baseline (Visit 1).

   However, if a history of ulcers is confirmed by the medical interview or previous medical record, Participants whose gastric ulcer scar or duodenal ulcer scar has disappeared may be included in the study.
3. Outpatient (including inpatient for examination)

Exclusion Criteria:

1. Participants who have received H.pylori eradication treatment
2. Participants who have either acute upper gastrointestinal bleeding, gastric ulcer [mucosal defect (with white coating including clot adherence) of 3 mm or larger in size], duodenal ulcer [mucosal defect (with white coating including clot adherence) of 3 mm or larger in size], acute gastric mucosal lesion (AGML), or acute duodenal mucosal lesion (ADML) on endoscopic examination at baseline (Visit 1).

   However, participants with gastric erosion or duodenal erosion may be included in the study.
3. Participants who have received or who are scheduled to undergo surgery which affects gastric acid secretion (ex, resection of upper gastrointestinal tract, vagotomy, etc)
4. Participants who cannot be treated with medicinal treatment (ex, perforation, pyloric stenosis or large hemorrhage, etc)
5. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders
6. Participants with hepatic or renal impairment receiving treatment with colchicines
7. Participants who have a history of hypersensitivity or allergy to TAK-438 (including its excipients), PPIs, penicillin antibiotics, macrolide antibiotics, or antitrichomonal agents
8. Participants with infectious mononucleosis
9. Participants with an organic disease of the brain or spinal cord

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate 4 weeks after completion of first-line therapy | 4-weeks post-dose (first-line therapy)
  The participants are judged to be H. pylori-negative or H. pylori-positive based on the 13C-Urea Breath Test.

SECONDARY OUTCOMES:
H. pylori eradication rate 4 weeks after completion of second-line therapy | 4-weeks post-dose (second-line therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (35):
- Japan (35):
  - Abiko-shi, Chiba
  - Kashiwa-shi, Chiba
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Ishikari-shi, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Marugame-shi, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Ebina-shi, Kanagawa
  - Yokohama, Kanagawa
  - Yatsushiro-shi, Kumamoto
  - Kyoto, Kyoto
  - Ōita, Oita Prefecture
  - Hirakata-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Takatsuki-shi, Osaka
  - Toyonaka-shi, Osaka
  - Saga, Saga-ken
  - Kumagaya-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Shizuoka, Shizuoka
  - Adachi-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Kokubunji-shi, Tokyo
  - Nishi-Tokyo-shi, Tokyo
  - Oota-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo

REFERENCES:
- [Derived] Murakami K, Sakurai Y, Shiino M, Funao N, Nishimura A, Asaka M. Vonoprazan, a novel potassium-competitive acid blocker, as a component of first-line and second-line triple therapy for Helicobacter pylori eradication: a phase III, randomised, double-blind study. Gut. 2016 Sep;65(9):1439-46. doi: 10.1136/gutjnl-2015-311304. Epub 2016 Mar 2. PMID 26935876